CLINICAL TRIAL: NCT07351877
Title: Exploring the Clinical Benefits of Precision Vibration on Neuromuscular Induction, Proprioceptive Gain, Functional Enhancement, and Pain Relief in Older Adults and and Stroke Survivors
Brief Title: Precision Vibration Therapy for Neuromuscular and Functional Improvement in Older Adults and Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC1130707-E
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Aging; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This project consists of two independent parallel sub-studies targeting different populations:
  1. older adults without stroke and
  2. stroke survivors (≥18 years, any age). Each sub-study uses a randomized parallel-group design comparing vibration therapy (upper or lower limb) versus conventional rehabilitation. The two populations will not be enrolled concurrently in the same study phase.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to participants' group allocation to reduce assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Older Adults (Conventional Rehabilitation) (Active Comparator): Older adults without stroke receive 60 minutes of conventional rehabilitation per session, including individualized strength, mobility, and balance training. Therapy duration is matched to the intervention group. Outcomes assessor is blinded.
  Interventions: Other: Conventional Rehabilitation
- Older Adults (Vibration Therapy on Upper or Lower Limb) (Experimental): Older adults without stroke receive 20 minutes of precision vibration therapy (applied to the upper or lower limb according to primary deficit) followed by 40 minutes of conventional rehabilitation per session. The total session time equals 60 minutes. Outcomes assessor is blinded.
  Interventions: Device: Precision Vibration Therapy
- Stroke Survivors (Conventional Rehabilitation) (Active Comparator): Stroke survivors (≥18 years) receive 60 minutes of conventional rehabilitation per session, including task-specific training, strengthening, and mobility exercises. Therapy duration is matched to the intervention group. Outcomes assessor is blinded.
  Interventions: Other: Conventional Rehabilitation
- Stroke Survivors (Vibration Therapy on Upper or Lower Limb) (Experimental): Stroke survivors receive 20 minutes of precision vibration therapy applied to the affected upper or lower limb followed by 40 minutes of conventional rehabilitation per session (total 60 minutes). Intervention aims to improve muscle strength, proprioception, and functional outcomes. Outcomes assessor is blinded.
  Interventions: Device: Precision Vibration Therapy

INTERVENTIONS:
Device: Precision Vibration Therapy — Precision vibration therapy applied to either the upper or lower limb, depending on participant's functional deficit. Each session includes 20 minutes of vibration followed by 40 minutes of conventional rehabilitation (total 60 minutes). The vibration device delivers controlled frequency and amplitude for neuromuscular activation, proprioceptive enhancement, and functional improvement.
  Arms: Older Adults (Vibration Therapy on Upper or Lower Limb); Stroke Survivors (Vibration Therapy on Upper or Lower Limb)
Other: Conventional Rehabilitation — Conventional rehabilitation therapy including task-specific training, strengthening, mobility, and balance exercises. Each session lasts 60 minutes. The therapy protocol is standardized across study sites and matched in duration and therapist contact time to the vibration therapy arms.
  Arms: Older Adults (Conventional Rehabilitation); Stroke Survivors (Conventional Rehabilitation)

SUMMARY:
To address muscle weakness, sensory degradation, functional decline, and pain caused by geriatric syndromes in older adults and stroke survivors, this project proposes a series of studies aimed at improving neuromuscular performance, muscle strength, proprioceptive gain, functional outcomes, and pain relief through the use of a precise vibration system.

In the first phase, a vibration exercise system will be implemented to recruit frail older adults and older adults with stroke for clinical trials. The goal is to verify the benefits of vibration intervention on limb muscle strength, proprioception, and movement function.

In the third phase, quantitative pain assessments and related scales will be used to evaluate chronic pain thresholds and affected regions in older adults and stroke survivors, and to validate the effectiveness of vibration intervention in alleviating their pain.

ELIGIBILITY:
Inclusion Criteria:

Older Adults:

* Meet two or more criteria of the Study of Osteoporotic Fractures (SOF) frailty index
* Willing to participate in the study and comply with all study procedures
* Able to wear and safely use the vibration device
* Normal cognitive function (Mini-Mental State Examination [MMSE] score ≥ 23)
* Presence of knee joint pain in the lower limbs

Stroke Survivors:

* Clinical diagnosis of ischemic or hemorrhagic stroke confirmed by a physician
* Clinically stable stroke condition (i.e., not in an acute or unstable phase)
* Brunnstrom stage ≥ III for the affected limb
* Cognitive ability sufficient to follow study procedures (MMSE score ≥ 23)
* Modified Ashworth Scale (MAS) score < 3 for the paretic limb
* Able to sit safely and participate in vibration or rehabilitation sessions for up to 60 minutes per visit
* Willing and able to comply with all study procedures and provide written informed consent

Exclusion Criteria:

Older Adults:

* Acute or chronic neurological injury involving the upper or lower limbs within the past 6 months
* Acute or chronic musculoskeletal injury involving the upper or lower limbs within the past 6 months
* History of surgery on the upper or lower limbs within the past 6 months

Stroke Survivors:

* Recurrent stroke during the current episode (i.e., acute re-stroke) or otherwise clinically unstable stroke presentation
* Markedly elevated spasticity preventing isolated voluntary movement of the target limb (MAS score ≥ 3)
* Hemianopsia or severe hemineglect that significantly interferes with task execution
* Concomitant vestibular or cerebellar disorders that severely impair motor performance
* Orthopedic or traumatic comorbidities causing significant pain or limiting safe participation during evaluation or intervention
* Cognitive impairment attributable to stroke that precludes effective communication or adherence to the study protocol
* Other neurological or psychiatric disorders judged likely to interfere with motor performance or study outcomes

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2027-12-18 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) Score | Baseline and Week 8 (end of intervention)
  The Fugl-Meyer Assessment evaluates motor recovery after stroke, including upper and lower extremity motor performance, coordination, and reflex activity. Higher scores indicate better motor function.
Motor Assessment Scale (MAS) Score | Baseline and Week 8 (end of intervention)
  The Motor Assessment Scale measures functional motor performance across multiple daily activities in stroke patients. Higher scores indicate better motor ability.
Maximal Voluntary Contraction (MVC) Force | Baseline and Week 8 (end of intervention)
  Maximal voluntary contraction of major lower-limb muscles will be measured using isometric dynamometry to assess muscle strength changes.
Muscle Force Stability | Baseline and Week 8 (end of intervention)
  Muscle force steadiness during submaximal contraction tasks will be quantified to evaluate neuromuscular control and stability.
Surface Electromyography (EMG) Activity | Baseline and Week 8 (end of intervention)
  Surface EMG recordings from target muscles will be used to analyze muscle activation patterns, coordination, and fatigue characteristics.
Pain Intensity (Visual Analog Scale, VAS) | Baseline and Week 8 (end of intervention)
  Pain intensity will be assessed using the 10-cm Visual Analog Scale (VAS), where higher scores indicate greater pain severity.
Functional Performance and Quality of Life | Baseline and Week 8 (end of intervention)
  Functional ability and perceived quality of life will be assessed using validated scales including the Barthel Index (BI), Instrumental Activities of Daily Living (IADL), and SF-36 Health Survey.
6-Minute Walk Test (6MWT) Distance | Baseline and Week 8 (end of intervention)
  The 6MWT measures functional endurance and walking capacity. Total distance walked in six minutes is recorded; longer distance indicates improved endurance.
10-Meter Walk Test (10MWT) Speed | Baseline and Week 8 (end of intervention)
  The 10MWT assesses gait speed and mobility. Average walking speed (m/s) over a 10-meter distance is calculated, with faster speeds indicating improved functional mobility.
30-Second Chair Stand Test Performance | Baseline and Week 8 (end of intervention)
  The 30-Second Chair Stand Test measures lower-limb strength and endurance by counting the number of full stands completed in 30 seconds. Higher counts indicate better performance.
Functional Reach Test Distance | Baseline and Week 8 (end of intervention)
  The Functional Reach Test assesses dynamic balance by measuring the maximum forward reach distance while maintaining a fixed base of support. Greater reach distance indicates better balance control.

SECONDARY OUTCOMES:
Minnesota Manual Dexterity Test (MMDT) Performance | Baseline and Week 8 (end of intervention)
  The Minnesota Manual Dexterity Test assesses manual dexterity and coordination of the upper limbs. Performance time (seconds) is recorded; shorter completion times indicate better dexterity.
Joint Proprioception (Active and Passive Position Sense) | Baseline and Week 8 (end of intervention)
  Measures active and passive joint position sense at upper and/or lower limb joints using standard proprioceptive testing procedures. Lower error angles indicate improved proprioceptive acuity.
Coordination Control (Bimanual Grip and Bilateral Ankle Coordination Tests) | Baseline and Week 8 (end of intervention)
  Coordination tests include bilateral grip control and bilateral ankle coordination tasks to evaluate interlimb coordination and control precision.
Barthel Index (BI) Score | Baseline and Week 8 (end of intervention)
  The Barthel Index assesses activities of daily living (ADL) independence, including feeding, bathing, dressing, mobility, and toileting. Higher scores indicate greater functional independence.
Wolf Motor Function Test (WMFT) Score | Baseline and Week 8 (end of intervention)
  The WMFT evaluates upper extremity motor function through timed and functional tasks. Lower time scores and higher functional ratings represent better motor performance.
Berg Balance Scale (BBS) Score | Baseline and Week 8 (end of intervention)
  The BBS assesses static and dynamic balance using 14 tasks. Total scores range from 0 to 56, with higher scores representing better balance.
Timed Up and Go (TUG) Test Performance | Baseline and Week 8 (end of intervention)
  The TUG test measures mobility and dynamic balance by recording the time taken to stand from a chair, walk 3 meters, turn, return, and sit. Shorter times indicate improved mobility.
Function (Spatiotemporal Parameters) | Baseline and Week 8 (end of intervention)
  Gait performance parameters (e.g., gait speed, stride length, cadence, and symmetry) will be assessed to evaluate locomotor function improvement.
Pain-Related Outcomes (BPI, PADT, PDI, NPRS) | Baseline and Week 8 (end of intervention)
  Pain characteristics and interference will be assessed using the Brief Pain Inventory (BPI), Pain Assessment and Documentation Tool (PADT), Pain Disability Index (PDI), and Numeric Pain Rating Scale (NPRS).
WOMAC Osteoarthritis Index | Baseline and Week 8 (end of intervention)
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will evaluate pain, stiffness, and physical function related to knee discomfort.
Quantitative Sensory Testing (QST) Results | Baseline and Week 8 (end of intervention)
  Quantitative sensory testing will be used to assess somatosensory function, including pain threshold and sensitivity.
Quality of Life (QOL and SF-36) | Baseline and Week 8 (end of intervention)
  Overall quality of life and health-related well-being will be assessed using the Quality of Life Questionnaire (QOL) and SF-36 Health Survey.

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Geriatrics and Welfare Research, National Health Research Institutes, Taipei, Taiwan